CLINICAL TRIAL: NCT03210753
Title: Study of Risk Factors and Genetic Association With Bortezomib-induced Peripheral Neuropathy in Multiple Myeloma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201610048RINA
Record Dates: First submitted 2017-07-02; First posted 2017-07-07 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Peripheral neuropathy; Subcutaneous injection; Bortezomib; Risk factors
MeSH Terms: conditions — Multiple Myeloma; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background and objective

The introduction of a proteasome inhibitor bortezomib has significantly improved response rates and overall survival in patients with multiple myeloma (MM), and it has soon become the cornerstone of treatment in both newly diagnosed and relapsed/refractory settings. However, the incidence of peripheral neuropathy related to bortezomib (BiPN) is unignorable and which becomes an obstacle during treatment with bortezomib, either alone or in combination. Until now, there are no consistent findings regarding the risk factors that may cause BiPN. There is either lack of large scale study of BiPN in Taiwan. This study aims to clarify risk factors of BiPN using retrospective analysis in a large cohort with longer observation period as well as the relations between BiPN and gene polymorphisms, and to compare different routes in the incidence of BiPN.

Methods

This is a retrospective cohort study with a sample size of about 400 MM patients treated ever with at least one full cycle of bortezomib in the institution. All the patients enrolled need to be adults (≧20 years ) with measurable M-component in either blood or urine. The investigators will perform a retrospective chart review to collect clinical data, including anti-MM and concomitant medications, to evaluate the incidence and severity of BiPN in this cohort, as well as any meaningful risk factors contributed to BiPN. The investigators also plan to perform genotyping for the possible genetic factors associated with development of BiPN.

Expected contributions

The successful collaboration between clinical hematologist-oncologist and biopharmaceutical researcher would result in the concrete evidence of efficacy and safety of bortezomib in Taiwanese patients with MM. The findings in this large cohort study will unveil the risk factors of BiPN, including the administration routes and ethnicity. As results, the investigators would be able to provide the precision medicine-based bortezomib treatment strategy to MM patients in Taiwan.

ELIGIBILITY:
Inclusion criteria

1. Age >20 years
2. Diagnosed with MM
3. Bortezomib new users (2006/4/1-2016/6/30)

Exclusion criteria

1. Varying on IV and SC administration
2. Receive bortezomib at other hospitals

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population from a medical center in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
peripheral neuropathy | 2006/4/1-2016/12/31
  identified the record of peripheral neuropathy, neuropathy, numbness, tingling, weakness symptoms by chart review

CONTACTS AND LOCATIONS:
Overall Officials: Huang Shang-Yi, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan